CLINICAL TRIAL: NCT01321073
Title: DelIVery for Pulmonary Arterial Hypertension (PAH) Clinical Study
Brief Title: DelIVery for Pulmonary Arterial Hypertension (PAH) & Continued Support Study
Acronym: DelIVery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Collaborators: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PAH-D
Record Dates: First submitted 2011-03-21; First posted 2011-03-23 (Estimated); Results first posted 2018-05-04 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-12

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Intervention Model Description: The study is observational and intended to provide ongoing support for the approximately 20 remaining subjects enrolled in the DelIVery for PAH Study including support of pump refills and system replacements. The study is expected to continue at the eight (8) remaining centers located in the United States that have current DelIVery for PAH study subjects enrolled.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DelIVery for Pulmonary Arterial Hypertension Single Arm (Experimental): All subjects were enrolled for implantation of the Model 10642 Implantable Intravascular Catheter used in combination with the SynchroMed II Implantable Infusion System (Model 8637) to deliver Remodulin Injection.
  Interventions: Device: Model 10642 Implantable Intravascular Catheter

INTERVENTIONS:
Device: Model 10642 Implantable Intravascular Catheter — This clinical study consists of the Model 10642 Implantable Intravascular Catheter used in combination with the SynchroMed II Implantable Infusion System (Model 8637) to deliver Remodulin Injection. This study will focus on the safety of delivery of Remodulin Injection in the treatment of patients with PAH who meet the approved Remodulin Injection indication, using the approved formulation, and approved intravenous route of administration.
  Other Names: Device: SynchroMed II Implantable Infusion System; Drug: Remodulin

SUMMARY:
The purpose of the DelIVery for PAH clinical study is to evaluate the safety of the Medtronic Model 10642 Implantable Intravascular Catheter when used with the Medtronic SynchroMed® II Implantable Infusion System to deliver Remodulin® (treprostinil) Injection.

As of June 2021, PMA approval of the Implantable System for Remodulin (ISR) is no longer being pursued and development and commercialization efforts have been halted. The approximately 30 subjects still implanted with the PIVoT system require a pathway for continued support. This protocol is amended and is designed to allow such ongoing support.

DETAILED DESCRIPTION:
Pulmonary arterial hypertension (PAH) is a severe, chronic syndrome affecting the small pulmonary arteries (blood vessels which carry blood from the heart to the lungs to pick up oxygen). At the time of the initiation of this study, no cure exists for this disease. Medtronic has developed a fully implantable, long term, intravenous infusion system, which has the potential to enhance patient convenience and ease of use, while reducing the opportunities for catheter-related infections and complication issues associated with currently used external delivery systems. The information gained from this study could provide evidence to support use on an implantable infusion system for the management of other disease states requiring chronic intravenous therapy. Additionally, information collected from this study may contribute to the design of new product(s)/therapy(ies) and/or instructions for use.

The purpose of this clinical study is to evaluate the safety profile of the Model 10642 Implantable Intravascular Catheter portion of the PAH Implantable Vasodilator Therapy (PIVoT) system. This study will focus on the safety of delivery of Remodulin Injection in the treatment of patients with PAH who meet the approved Remodulin Injection indication, using the approved formulation, and approved intravenous route of administration.

The Model 10642 Implantable Intravascular Catheter being used in this study is investigational, meaning it has not been approved by the FDA to be safe. The Model 10642 Catheter is different from other commercially available drug delivery catheters because the Model 10642 Catheter tube has a one-way valve designed to allow the medication to flow out but keep blood from flowing back into the catheter tube. The Model 10642 Catheter is reinforced to prevent kinking and crushing, which could interrupt the flow of medication.

Remodulin Injection is a Food and Drug Administration (FDA) approved drug for the intravenous and subcutaneous treatment of PAH.

The SynchroMed II Implantable Infusion System is approved by the FDA to deliver specific drugs in patients who have chronic pain, need management of severe spasticity, and for cancer treatment but has not been approved to deliver Remodulin Injection in patients with PAH.

There is also a Catheter Imaging Sub-Study that is being done to measure the shape change of the Model 10642 Implantable Intravascular Catheter during a given set of patient positions through the use of x-ray imaging. This data will help us develop more clinically realistic bench tests and simulations that better mimic the challenges experienced by an implanted catheter. This Catheter Imaging Sub-Study will be conducted at up to seven centers and will enroll up to forty patients that are currently enrolled in the DelIVery for PAH clinical study and are at least three months post-implant of their current catheter and pump.

ELIGIBILITY:
Inclusion Criteria:

* Patient is currently enrolled in the DelIVery for PAH Study (G100017)
* The physician and patient determine that continued use of the PIVoT system is medically advisable
* Patient is willing to sign and date the Patient Informed Consent Form

Exclusion Criteria:

- N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2013-06 (Actual); Study Completion 2032-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: DelIVery for PAH Clinical Research Specialist, Study Chair — Medtronic
Locations (8):
- United States (8):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - VA Greater Los Angeles Healthcare System, Los Angeles, California
  - AdventHealth Orlando, Orlando, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Aurora St. Lukes Medical Center, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Waxman AB, McElderry HT, Gomberg-Maitland M, Burke MC, Ross EL, Bersohn MM, Pangarkar SS, Tarver JH, Zwicke DL, Feldman JP, Chakinala MM, Frantz RP, Thompson GB, Torres F, Rauck RL, Clagg K, Durst L, Li P, Morris M, Southall KL, Peterson L, Bourge RC. Totally Implantable IV Treprostinil Therapy in Pulmonary Hypertension Assessment of the Implantation Procedure. Chest. 2017 Dec;152(6):1128-1134. doi: 10.1016/j.chest.2017.04.188. Epub 2017 Jun 3. PMID 28583617
- [Background] Gomberg-Maitland M, Bourge RC, Shapiro SM, Tarver JH 3rd, Zwicke DL, Feldman JP, Chakinala MM, Frantz RP, Torres F, Bag R, Murphy JA, Lautenbach AA, Morris M, Peterson L, Waxman AB. Long-term results of the DelIVery for Pulmonary Arterial Hypertension trial. Pulm Circ. 2019 Nov 5;9(4):2045894019878615. doi: 10.1177/2045894019878615. eCollection 2019 Oct-Dec. PMID 31723407
- [Background] Shapiro S, Bourge RC, Pozella P, Harris DF, Borg EH, Nelsen AC. Implantable system for treprostinil: a real-world patient experience study. Pulm Circ. 2020 Apr 22;10(2):2045894020907881. doi: 10.1177/2045894020907881. eCollection 2020 Apr-Jun. PMID 32363029
- [Background] Feldman JP, Gomberg-Maitland M, Shapiro SM, Lautenbach AA, Morris M, Murphy JA, Waxman AB, Bourge RC. Implantable system for treprostinil and lung transplantation: case series from delivery for pulmonary arterial hypertension study. Pulm Circ. 2021 Mar 2;11(1):2045894021999290. doi: 10.1177/2045894021999290. eCollection 2021 Jan-Mar. PMID 33738097
- [Result] Bourge RC, Waxman AB, Gomberg-Maitland M, Shapiro SM, Tarver JH 3rd, Zwicke DL, Feldman JP, Chakinala MM, Frantz RP, Torres F, Cerkvenik J, Morris M, Thalin M, Peterson L, Rubin LJ. Treprostinil Administered to Treat Pulmonary Arterial Hypertension Using a Fully Implantable Programmable Intravascular Delivery System: Results of the DelIVery for PAH Trial. Chest. 2016 Jul;150(1):27-34. doi: 10.1016/j.chest.2015.11.005. Epub 2016 Jan 13. PMID 27396777

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DelIVery for Pulmonary Arterial Hypertension Single Arm
Started | 64
Completed | 57
Not Completed | 7
Not completed — Did not attempt implant | 4
Not completed — Death | 3

BASELINE CHARACTERISTICS:
Population: All patients attempting implant
Arm/Group | DelIVery for Pulmonary Arterial Hypertension Single Arm
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.1 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2
  Black or African American | 3
  Hispanic or Latino | 8
  White or Caucasian | 47
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Rate of Catheter-related Complications Per 1000 Patient Days
Description: A complication is an adverse event that required an invasive intervention. Complications related to the implanted catheter are counted. In addition, because pneumothoraxes are counted as part of the endpoint.
Time Frame: Implant to 2 years
Population: All days of follow-up for implanted patients
Measure: Number; unit: complications per 1000 patient-days
Units Other Than Participants: Patient days
Arm/Group | DelIVery for Pulmonary Arterial Hypertension Single Arm
Number analyzed (Participants) | 60
Number analyzed (Patient days) | 22013
complications per 1000 patient-days | 0.27
Statistical Analysis 1: Comparison: DelIVery for Pulmonary Arterial Hypertension Single Arm; The rate of catheter-related complications per 1000 patient-days was compared to a pre-specified value of 2.5 / 1000 days. This was calculated based on published complication rates in PAH that included central venous catheter systemic bloodstream infections (0.43-1.13), site infections (0.26-0.87), and complications from catheter thrombosis, mechanical dysfunction, or catheter dislocation in the general central venous catheter population (0.36-0.51). The sum of the upper rates is 2.5; Test type: Superiority; p < 0.0001, 1-sample exact test for Poisson rate

ADVERSE EVENTS:
Time Frame: Implant to 24 months
Description: An adverse event is any untoward medical occurrence in a subject. Serious Adverse Events include adverse events that result in death, require either inpatient hospitalization or the prolongation of hospitalization, are life-threatening, a persistent or significant disability/incapacity or a congenital anomaly/birth defect. Other important medical events, based upon medical judgment, may also be considered serious if a trial participants' health is at risk and intervention is required.
Groups:
- Single Arm: All subjects were enrolled for implantation of the Model 10642 Implantable Intravascular Catheter used in combination with the SynchroMed II Implantable Infusion System (Model 8637) to deliver Remodulin Injection.
  Model 10642 Implantable Intravascular Catheter: This clinical study consists of the Model 10642 Implantable Intravascular Catheter used in combination with the SynchroMed II Implantable Infusion System (Model 8637) to deliver Remodulin Injection. This study will focus on the safety of delivery of Remodulin Injection in the treatment of patients with PAH who meet the approved Remodulin Injection indication, using the approved formulation, and approved intravenous route of administration.
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 3/60
Serious Adverse Events (participants affected / at risk) | 29/60
Other Adverse Events (participants affected / at risk) | 57/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=60)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Autoimmune thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Atrial flutter (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Right ventricular failure (Cardiac disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Device damage (General disorders) | 1 (1)
Device dislocation (General disorders) | 2 (3)
Immediate post-injection reaction (General disorders) | 3 (3)
Implant site effusion (General disorders) | 1 (1)
Injection site reaction (General disorders) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Implant site infection (Infections and infestations) | 1 (1)
Lobar pneumonia (Infections and infestations) | 1 (1)
Lyme disease (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (2)
Pneumonia legionella (Infections and infestations) | 1 (1)
Rhinovirus infection (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Postoperative fever (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 2 (2)
Gout (Metabolism and nutrition disorders) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Renal failure chronic (Renal and urinary disorders) | 1 (1)
Endometriosis (Reproductive system and breast disorders) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (2)
Venous stenosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=60)
Abdominal pain (Gastrointestinal disorders) | 6 (6)
Constipation (Gastrointestinal disorders) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 5 (5)
Nausea (Gastrointestinal disorders) | 11 (11)
Vomiting (Gastrointestinal disorders) | 4 (4)
Fatigue (General disorders) | 6 (6)
Implant site bruising (General disorders) | 10 (10)
Implant site pain (General disorders) | 51 (54)
Injection site pain (General disorders) | 4 (4)
Injection site reaction (General disorders) | 9 (10)
Nasopharyngitis (Infections and infestations) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 17 (21)
Procedural vomiting (Injury, poisoning and procedural complications) | 4 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (7)
Dizziness (Nervous system disorders) | 7 (7)
Headache (Nervous system disorders) | 8 (10)
Insomnia (Psychiatric disorders) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 (16)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 8 (9)
Flushing (Vascular disorders) | 5 (5)
Hypotension (Vascular disorders) | 9 (9)

LIMITATIONS AND CAVEATS:
Results are through June, 2013 when 22,000 patient days of implant had been accumulated. This was the pre-specified primary analysis time for the study. The study continued past this point.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less